CLINICAL TRIAL: NCT05513092
Title: Role of Placenta Accreta Index in Predicting Conservative Surgery for Placenta Accreta Spectrum
Brief Title: Placenta Accreta Index Score in Placenta Accreta Spectrum
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: 10544
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Placenta Accreta, Third Trimester
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: placenta accreta index score — role of placenta accreta index score in prediction of conservative surgery for placenta placenta accreta spectrum

SUMMARY:
role of placenta accreta index score in prediction of conservative surgery for placenta placenta accreta spectrum

DETAILED DESCRIPTION:
in this study ,we will recruit 60 cases diagnosed placenta previa accreta by 2D ultrasound and Doppler then patients will have 3D Doppler to calculate placenta accreta index score according to agarawl et al criteria , patients will have cs accroding to our hospital protocol "Al demerdash maternity hospital ,Ainshams university" .Intraoperative findings will be noticed ,postoperative histopathological examination may br needed in cases of cs hystrectomy ,placenta accreta index score will be compared to intra and postoperative findings , patients will be followed up for two weeks after delivery for any postoperative complication

ELIGIBILITY:
Inclusion Criteria:

* • Pregnant women above 28 weeks gestation by 1st trimesteric U/S,2nd trimesteric U/S or sure reliable dates; diagnosed as placenta previa by 2D ultrasound, Doppler on placental bed.

  * Patients who have done one or more cesarean sections

Exclusion Criteria:

* Patients who refuse to participate in our study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: • Pregnant women above 28 weeks gestation by 1st trimesteric U/S,2nd trimesteric U/S or sure reliable dates; diagnosed as placenta previa by 2D ultrasound, Doppler on placental bed.
  Patients who have done one or more cesarean sections
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of PAS index score in prediction of conservative surgery | 2022 to 2024

SECONDARY OUTCOMES:
Intraoperative blood loss | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mamdouh, Study Director — Ainshams university
Locations (1):
- Ainshams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided